CLINICAL TRIAL: NCT01013363
Title: Music as an Auxiliary Analgesic and Anxiolytic During First Trimester Abortion
Brief Title: The Use of Music for Pain and Anxiety Control During Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Family Planning Fellowship (Other)
Responsible Party: Principal Investigator, Paula Castano, Assistant Clinical Professor, Columbia University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAE0439
Record Dates: First submitted 2009-11-06; First posted 2009-11-13 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2012-11

CONDITIONS: Pain; Anxiety
Keywords: abortion; first trimester; suction aspiration; vacuum aspiration; music; anesthesia; analgesia; anxiolytic; pain; anxiety; blood pressure; heart rate; satisfaction
MeSH Terms: conditions — Pain; Anxiety Disorders; Agnosia; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No music (No Intervention): Participants will not use the digital music player during their procedure.
- Music (Experimental): Participants will use the digital music player during their procedure.
  Interventions: Other: iPod Nano digital music player

INTERVENTIONS:
Other: iPod Nano digital music player — Digital music player pre-loaded with 10 playlists to be used intra-operatively by the participant randomized to the intervention group.
  Arms: Music

SUMMARY:
Most first trimester abortions are performed under local anesthesia using either manual or electric vacuum suction aspiration. The majority of women undergoing these procedures experience some amount of pain and anxiety. The investigators seek to understand if the provision of music during first trimester abortion will reduce pain and anxiety associated with this procedure. This study will involve the use of music during first trimester abortion as an additional method of pain and anxiety control. The investigators will recruit women seeking a first trimester suction aspiration procedure primarily for elective pregnancy termination or for other related indications such as an abnormal pregnancy, inevitable abortion, or retained products of conception. Participation will be voluntary and include informed consent. Recruited women will be divided into two groups: control group (no music) and intervention (music) group. All subjects will receive routine care and standard pain control measures, including local anesthesia, during their procedure. Those assigned to the intervention group will receive a portable digital music player (iPOD™ Nano) with headphones to listen to during their procedure. All subjects will complete preoperative and postoperative pain and anxiety questionnaires in addition to a patient satisfaction survey at the end of their visit. The provider will also assess and record the subject's pain experienced during the procedure. The investigators will also measure preoperative and postoperative vital signs on all participants. Subjects will be compensated for their time and study participation will not affect any care received at the clinic. Upon completion of their visit, there will be no additional followup for this study.

DETAILED DESCRIPTION:
Nearly 90% of abortions occur during the first trimester and a majority of these are performed by suction curettage in an outpatient setting using local anesthesia (Grimes, 2007; Lichtenberg, 2001). When only local anesthesia is used, 97% of women experience pain, and anxiety level is a positive predictor of pain during abortion (Bélanger, 1989). Although general anesthesia offers better agents for anxiety and pain management, this route is less commonly used because of prohibitive costs and potential complications (Grimes, 2007). Because many first trimester abortion providers utilize local anesthesia as primary pain management during the procedure, multiple agents and techniques have been investigated to supplement or enhance the effects of the local anesthetic. Investigated methods include time delay between paracervical block administration and cervical dilation, intrauterine lidocaine infusion, and various combinations of inhaled, oral, and intravenous analgesics and anxiolytics. Additionally, complementary and alternative regimens such as relaxation, distraction, hypnosis, and aromatherapy have also been evaluated as auxiliary analgesics and anxiolytics during first trimester abortion. Despite these attempts to improve the anxiety and pain associated with abortion under local anesthesia, the results and efficacy of these methods is variable and inconsistent.

Music therapy is classified as a cognitive-behavioral intervention that helps patients by providing them with a greater sense of self-control in assessing and managing pain (AHCPR, 1992). In 1992, recommendations by the Agency for Healthcare Research and Quality included music as one type of cognitive-behavioral intervention for pain management (AHCPR, 1992). The exact mechanism as to how music impacts pain sensory systems has not been fully elucidated, but it is thought to engage specific brain functions involved in memory, learning, and multiple motivational and emotional states (Nilsson, 2008). As the most influential theory on the nature of pain, the Gate Control Theory hypothesizes that cognitive-behavioral interventions work by closing the gate of nerve fibers that transmit ascending sensory information to the brain while concurrently modulating input from inhibitory systems and psychological factors, the sum of which leads to a reduction in the pain experience (Tse, 2005; Sendelbach, 2006). The Gate Control Theory posits that music acts as a distracter, diverting attention away from a noxious stimulus by redirecting a person's attention or by involving the individual in a distracting task (Tse, 2005).

The role of music as an auxiliary analgesic and anxiolytic has been evaluated in such outpatient procedures as colonoscopy, laceration repair, dental work, lithotripsy, nasal surgery, breast biopsy, and colposcopy (Chan, 2003). In addition to other nonpharmacologic approaches to pain management such as relaxation, distraction, and guided imagery, musical interventions have demonstrated favorable effects upon pain, anxiety, wound healing, and recovery among patients in the peri-operative setting (Laurion, 2003). Physiological parameters such as heart rate, blood pressure, and stress hormone levels improve under the influence of music (Leardi, 2007). A Cochrane Collaboration review on the use of music for pain relief found that music reduced pain intensity levels but recommended that music not be used for primary pain control (Cepeda, 2006). The authors also concluded that the impact of music on anxiety has not yet been determined and needs to be further investigated. Given music's demonstrated benefits as an auxiliary analgesic and anxiolytic in multiple operative settings, its role in the abortion setting deserves further examination. The objective of this study is to evaluate the role of music as an alternative agent for pain and anxiety management during first trimester abortion.

A systematic review of 42 randomized controlled trials evaluated the effects of music in multiple peri-operative settings and found that the intervention had positive effects in reducing patient pain and anxiety in approximately half of the reviewed studies (Nilsson, 2008). Many included trials were noted to be of "insufficient quality" and a meta-analysis could not be performed due to variation in the types of music used, the duration of listening time, and procedures investigated. Furthermore, some studies used non-validated questionnaires and had other methodological limitations. Nonetheless, the author concluded that peri-operative musical interventions are easy to implement and effective in reducing patient pain, anxiety, and stress (Nilsson, 2008).

A 2006 Cochrane Collaboration review examined the effect of music on acute and chronic pain in 51 randomized controlled trials. They calculated the mean difference in pain intensity levels, percentage of patients with at least 50% pain relief, and opioid requirements among 3663 subjects. The authors concluded that listening to music reduced pain intensity levels and opioid requirements but that the magnitude of these benefits is small with uncertain clinical significance (Cepeda, 2006). Although the pooled results indicated statistical significance in the reduction of post-operative pain intensity levels, the authors stated that the role of music in pain relief warrants further investigation as does its role as a potential anxiolytic. As musical interventions have not been shown to have adverse effects, it is worth pursuing this nonpharmacologic agent as a supplemental resource for patients undergoing medical procedures such as first trimester abortion.

Only one study, published in 1975, has examined music as an auxiliary analgesic during first trimester abortion. This was a randomized controlled trial of 144 patients divided into 3 groups who all received oral diazepam and a paracervical block with mepivacaine in addition to 1) no further anesthesia, 2) self-administered methoxyflurane, or 3) music via stereophonic headphones. Patients who listened to music during suction curettage reported less tension and less pain (Shapiro, 1975). Although this study showed a beneficial effect of music, its findings are limited by poor study descriptors of patient characteristics, an unspecified randomization procedure, and lack of appropriate statistical analysis. A non-validated pain questionnaire was utilized and there is minimal description of procedural methods, the intervention, and results. Given these limitations, its results may not be applicable by current randomized trial guidelines. Nonetheless, this is the only published study to examine the use music as an auxiliary analgesic during first trimester abortion.

Because pain perception is also thought to be highly associated with comorbid conditions such as depression, anxiety, and substance abuse, the pain experience may influence overall satisfaction outcomes related to a specific event (Guzeldemir, 2008; Bair, 2007). The baseline presence of any of these conditions may impact one's response to pain management, anxiety status, and satisfaction associated with a procedure. In addition to overall satisfaction, we will assess for these comorbid conditions in our study.

Today, music has become very portable in the form of digital music players such as the iPOD™. With 25% of Americans and 51% of American adolescents owning one of these devices, music is a familiar part of many lives (Pew, 2006). Pain studies evaluating musical interventions as auxiliary analgesia have used various types of music via different delivery systems (i.e. cassette/CD player with headphones, loudspeakers, live music by a music therapist) in different settings. Many of these trials have utilized self-selection of music and have included a variety of musical genres, specific sounds, white noise, and vocal suggestions. Although some studies indicate that slow and non-lyrical music of the patient's choice for at least 30 minutes at 60 decibel volume is ideal for optimal pain relief and relaxation, it is not known if these factors directly influence music's impact in reducing pain and anxiety (Nilsson, 2008).

Additionally, there is mixed evidence on the role of patient choice in music selection and whether this affects the amount of pain or anxiety experienced. While some studies have advocated the use of self-selected music to enhance pain and anxiety reduction (Hekmat, 1993; Lee, 2004), the previously mentioned Cochrane review found that the decline in pain intensity was similar among patients whether or not the music was self-selected (Cepeda, 2006).

Given the data on music's potential ability to positively influence surgical experiences, we believe that music as an auxiliary method of anxiety and pain management in first trimester abortion warrants further investigation. The proposed study will evaluate music's impact on anxiety and pain experienced during first trimester abortion performed with local anesthesia and how this might influence overall satisfaction experienced with the procedure. Given that 50% of women who had abortions in 2005 were less than 25 years old (Gamble, 2008) and that this younger age group likely has increased familiarity with portable digital music players, this patient population may benefit from music as an auxiliary analgesic and anxiolytic during pregnancy termination. This research has the potential to expand the arsenal of low-cost, safe, and effective analgesics and anxiolytics available for surgical abortion, a commonly performed procedure across the United States and worldwide. The addition of music to first trimester abortion under local anesthesia provides an opportunity to improve the pain and anxiety associated with this procedure, especially given that many women of reproductive age utilize personal digital music players and may welcome this auxiliary analgesic and anxiolytic to their experience.

The proposed study will be a randomized controlled trial to evaluate the hypothesis that intraoperative music reduces patient anxiety and pain during first trimester abortion. We will examine the role of music as an auxiliary analgesic and anxiolytic in conjunction with a standard pain control regimen used in first trimester suction aspiration procedures consisting of preoperative oral ibuprofen and local anesthesia using a 1% lidocaine paracervical block. Participants will be randomized in a 1:1 ratio to the control and intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Viable or non-viable intrauterine pregnancy less than or equal to 14 weeks gestational age (including women with an abnormal pregnancy, inevitable abortion, or retained products of conception)
* Ability to read and speak English or Spanish
* Willingness to participate in the randomized trial

Exclusion Criteria:

* Hearing or visual impairment
* Allergy to ibuprofen or lidocaine

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Pain and anxiety experienced during first trimester abortion. | 1 day. Outcome measured immediately after procedure without additional follow-up.

SECONDARY OUTCOMES:
Heart rate and blood pressure changes. | Measured before and after procedure.
Overall patient satisfaction. | Assessed immediately after procedure.
Provider assessment of patient's pain. | Assessed immediately after procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Paula M Castano, MD, MPH, Principal Investigator — Columbia University; Jacqueline M Guerrero, MD, Study Director — Columbia University
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Result] Guerrero JM, Castano PM, Schmidt EO, Rosario L, Westhoff CL. Music as an auxiliary analgesic during first trimester surgical abortion: a randomized controlled trial. Contraception. 2012 Aug;86(2):157-62. doi: 10.1016/j.contraception.2011.11.017. Epub 2012 Jan 10. PMID 22240180
- [Derived] Oviedo JD, Ohly NT, Guerrero JM, Castano PM. Factors associated with participant and provider pain rating during office-based first-trimester vacuum aspiration. Contraception. 2018 Jun;97(6):497-499. doi: 10.1016/j.contraception.2018.01.001. Epub 2018 Jan 6. PMID 29317229